CLINICAL TRIAL: NCT02775084
Title: Nutritional Intervention to Test Effect on Healthy Human T Cell Function
Brief Title: Fish Oil T Cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB2015-0691
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Muscle Strength; Cognitive Function
Keywords: n-3; Polyunsaturated; Fatty acids; Antigens; Cognition; CD4
MeSH Terms: interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Fish Oil (Experimental): 8 grams fish oil
  Interventions: Dietary Supplement: Fish Oil
- Olive Oil (Placebo Comparator): 8 grams olive oil
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — 4 capsules twice daily with food for 6 weeks
  Arms: Healthy Fish Oil
Dietary Supplement: Olive Oil — 4 capsules twice daily with food for 6 weeks
  Arms: Olive Oil

SUMMARY:
The purpose of the study is to examine the effect of dietary n-3 polyunsaturated fatty acid supplementation on subjects' pan CD4+ T cell function, cognition, and muscle function. Half of the participants will receive fish oil, while the other half will receive a placebo (olive oil).

DETAILED DESCRIPTION:
Generalized inflammation has been consistently associated with aging and metabolic diseases, often characterized by reduced muscle and cognitive function. Although much of the aging-associated inflammation has been attributed to chronic activation of the innate host defense system, activated CD4+ T cells have been shown to contribute directly to the pathogenesis of several other inflammatory diseases. In humans, dietary n-3 polyunsaturated fatty acids (PUFA), particularly docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), have anti-inflammatory properties and reduce disease symptoms, in part, through suppression of CD4+ T cell activation. Therefore, the Researchers' overall hypothesis is that dietary supplementation with DHA and EPA in humans will ameliorate inflammatory symptoms, in part, by suppressing CD4+ T cell activation, positively affecting muscle and cognitive function.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male or female according to the investigator/appointed staff judgment
2. 55 years and older
3. Stable body weight for the past 3 months (< 5% change)

Exclusion criteria:

1. History of cardiovascular disease
2. Metabolic diseases, including hepatic or renal disorders
3. Presence of acute illness or metabolically unstable chronic illness (including diagnosis of Insulin Dependent Diabetes Mellitus)
4. Unwilling to stop taking nutritional supplements containing proteins or free amino acids within 5 days of the first study day until study completion
5. Participated in a nutritional supplement study program within the past 4 weeks
6. Any other condition according to the PI or nurse that would interfere with the study or safety of the subject or influence the results
7. Daily use of supplements containing > 1000 mg EPA+DHA 3 months prior to the first test day
8. Known hypersensitivity to fish and/or shellfish, Swanson EFAs Super EPA Fish oil or any of its ingredients, Swanson EFAs Certified Organic Extra Virgin Olive oil or any of its ingredients
9. Presence of fever within the last 3 days
10. Failure to give informed consent
11. (Possible) Pregnancy
12. Unwilling to comply with any other rules set forth in the Informed Consent Form

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in function of of lipid rafts in immune cell membranes due to dietary polyunsaturated fatty acids supplementation | one time on baseline, day 21 and day 42
  one blood draw on each study visit

SECONDARY OUTCOMES:
Fatty acid metabolism | one time on baseline, day 21 and day 42
  One blood draw on each study visit
Skeletal muscle strength of hand | 30 minutes on baseline, day 21 and day 42
  Measurement of hand grip strength
Skeletal muscle strength of leg | 30 minutes on baseline, day 21 and day 42
  Measurement of muscle strength of leg using kin-com machine
Body Composition | 15 minutes on baseline, day 21 and day 42
  Body composition as measured by Dual-Energy X-ray Absorptiometry
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  A fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Diet recall | on baseline and change from day 21 and day 42
  The subject is asked to recall in detail all the food and drink consumed during the 24 hours prior to the test day.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT) | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  A word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in attention and executive functions as measured by Trail Making Test (TMT) | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Group differences in learning and memory as measured by Digit Span | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  Recall of numbers in the same order (Digit Forward) and in reverse order (Digit Backward). Measures auditory attention and verbal working memory.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  Assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Executive Function-Adolescent/Adult Sensory Profile (ASP) | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  A standardized self-questionnaire that generates an individualized profile of sensory processing across four quadrants: low registration, sensation seeking, sensory sensitivity, and sensation avoiding.
Group differences in attention and executive functions as measured by Brief-A | Postabsorptive state during 1 hours and change after feeding on baseline and change from day 21 and day 42
  A standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No